CLINICAL TRIAL: NCT02542449
Title: Placebo Controlled, Randomized, Single Blinded Trial on the Effects of Greenselect Phytosome® on Weight Maintenance in Obese Women After a 3-month Weight Loss Intervention
Brief Title: Effects of Greenselect Phytosome® on Weight Maintenance After Weight Loss in Obese Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19A301_2013
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
Keywords: Green tea; weight maintenance; obesity; fat mass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Globes® (Active Comparator): Partecipants received twice a day for 3 months Globes® (Pharmextracta, Pontenure, Piacenza, Italy) formulated to be enteric-coated and containing 150 mg/dose of Greenselect Phytosome® and pure piperine (15 mg/dose) from Piper nigrum L.
  Interventions: Dietary Supplement: Globes®
- Placebo (Placebo Comparator): Partecipants received twice a day for 3 months placebo (undistinguishable from Globes in terms of size, shape, taste, odor, primary and secondary packaging).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Globes® — At the end of a 3-month lifestyle intervention, all participants received twice a day for 3 months Globes® and attended a monthly clinical visit during the supplementation period and 3 months after the end of supplementation.
  Arms: Globes®
Dietary Supplement: Placebo — At the end of a 3-month lifestyle intervention, all participants received twice a day for 3 months placebo and attended a monthly clinical visit during the supplementation period and 3 months after the end of supplementation.
  Arms: Placebo

SUMMARY:
This study evaluates whether supplementations with a highly bioavailable green tea extract may help obese women to counteract weight regain after a 3-month weight loss intervention.

DETAILED DESCRIPTION:
Most obese subjects regain weight after weight loss due to compensatory adaptations finalized to maintain stable body energy stores. In lean or obese individuals, maintenance of a 10% or greater reduction in body weight is associated with a decline in 24-hour energy expenditure of approximately 20%-25%. The restraint of the energy expenditure decline during dieting by green tea (GT) preparations should be a useful strategy to facilitate weight maintenance. To increase absorption of GT, the investigators used a formulation with phospholipids (Greenselect Phytosome® ) added with piperine, a thermogenic agent and a booster of absorption for various phenolics.

At the end of a 3-month lifestyle intervention, all patients giving written informed consent were randomly assigned to two groups for the weight-maintenance phase: 20 of them were supplemented twice a day for 3 months with a dietary supplement (Globes®, Pharmextracta, Pontenure, Piacenza, Italy) and 20 with placebo.Women were blind to the supplementation throughout the whole trial. All women attended a monthly clinical visit during the supplementation period and 3 months after the end of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* ≥18 years of age
* body mass index (BMI) ≥ 30 kg/m2
* a sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

* breast feeding or pregnancy
* history of cardiovascular or cerebrovascular events
* uncontrolled hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
change in body weight from baseline to 12 weeks of supplementation | baseline and 12 weeks of supplementation

SECONDARY OUTCOMES:
change in body weight from baseline to 4 weeks of supplementation | baseline and 4 weeks of supplementation
change in body weight from 4 weeks to 8 weeks of supplementation | 4 weeks and 8 weeks of supplementation
change in body weight from 8 weeks to 12 weeks of supplementation | 8 weeks and 12 weeks of supplementation
change in body weight from 12 weeks of supplementation to 3 months after discontinuation of supplementation | 12 weeks of supplementation and 3 months after discontinuation of supplementation
change in waist circumference from baseline to 12 weeks of supplementation | baseline and 12 weeks of supplementation
change in waist circumference from baseline to 4 weeks of supplementation | baseline and 4 weeks of supplementation
change in waist circumference from 4 weeks to 8 weeks of supplementation | 4 weeks and 8 weeks of supplementation
change in waist circumference from 8 weeks to 12 weeks of supplementation | 8 weeks and 12 weeks of supplementation
change in waist circumference from 12 weeks of supplementation to 3 months after discontinuation of supplementation | 12 weeks of supplementation and 3 months after discontinuation of supplementation
change in body composition from baselineto 12 weeks of supplementation | baseline and 12 weeks of supplementation
  Body composition was measured using a body composition analyzer with joined function of body fat analysis (Biki 300, Jawon Medical, Korea)
change in blood pressure from baseline to 12 weeks of supplementation | baseline and 12 weeks of supplementation
change in heart rate from baseline to 12 weeks of supplementation | baseline and 12 weeks of supplementation
change in body composition from baseline to 4 weeks of supplementation | baseline and 4 weeks of supplementation
  Body composition was measured using a body composition analyzer with joined function of body fat analysis (Biki 300, Jawon Medical, Korea)
change in blood pressure from baseline to 4 weeks of supplementation | baseline and 4 weeks of supplementation
change in heart rate from baseline to 4 weeks of supplementation | baseline and 4 weeks of supplementation
change in body composition from 4 weeks to 8 weeks of supplementation | 4 weeks and 8 weeks of supplementation
  Body composition was measured using a body composition analyzer with joined function of body fat analysis (Biki 300, Jawon Medical, Korea)
change in blood pressure from 4 weeks to 8 weeks of supplementation | 4 weeks and 8 weeks of supplementation
change in heart rate from 4 weeks to 8 weeks of supplementation | 4 weeks and 8 weeks of supplementation
change in body composition from 8 weeks to 12 weeks of supplementation | 8 weeks and 12 weeks of supplementation
  Body composition was measured using a body composition analyzer with joined function of body fat analysis (Biki 300, Jawon Medical, Korea)
change in blood pressure from 8 weeks to 12 weeks of supplementation | 8 weeks and 12 weeks of supplementation
change in heart rate from 8 weeks to 12 weeks of supplementation | 8 weeks and 12 weeks of supplementation
change in body composition from 12 weeks of supplementation to 3 months after discontinuation of supplementation | 12 weeks of supplementation and 3 months after discontinuation of supplementation
  Body composition was measured using a body composition analyzer with joined function of body fat analysis (Biki 300, Jawon Medical, Korea)
change in blood pressure from 12 weeks of supplementation to 3 months after discontinuation of supplementation | 12 weeks of supplementation and 3 months after discontinuation of supplementation
change in heart rate from 12 weeks of supplementation to 3 months after discontinuation of supplementation | 12 weeks of supplementation and 3 months after discontinuation of supplementation
the proportion of women with ≥ 5% weight loss | at 4 weeks of supplementation
the proportion of women with ≥ 5% weight loss | at 8 weeks of supplementation
the proportion of women with ≥ 5% weight loss | at 12 weeks of supplementation
the proportion of women with ≥ 5% weight loss | 3 months after discontinuation of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Invitti, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, Milano, Italy

REFERENCES:
- [Background] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981
- [Background] Hursel R, Westerterp-Plantenga MS. Catechin- and caffeine-rich teas for control of body weight in humans. Am J Clin Nutr. 2013 Dec;98(6 Suppl):1682S-1693S. doi: 10.3945/ajcn.113.058396. Epub 2013 Oct 30. PMID 24172301
- [Background] Jurgens TM, Whelan AM, Killian L, Doucette S, Kirk S, Foy E. Green tea for weight loss and weight maintenance in overweight or obese adults. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD008650. doi: 10.1002/14651858.CD008650.pub2. PMID 23235664
- [Background] Di Pierro F, Menghi AB, Barreca A, Lucarelli M, Calandrelli A. Greenselect Phytosome as an adjunct to a low-calorie diet for treatment of obesity: a clinical trial. Altern Med Rev. 2009 Jun;14(2):154-60. PMID 19594224
- [Background] Lambert JD, Hong J, Kim DH, Mishin VM, Yang CS. Piperine enhances the bioavailability of the tea polyphenol (-)-epigallocatechin-3-gallate in mice. J Nutr. 2004 Aug;134(8):1948-52. doi: 10.1093/jn/134.8.1948. PMID 15284381
- [Background] Dulloo AG, Duret C, Rohrer D, Girardier L, Mensi N, Fathi M, Chantre P, Vandermander J. Efficacy of a green tea extract rich in catechin polyphenols and caffeine in increasing 24-h energy expenditure and fat oxidation in humans. Am J Clin Nutr. 1999 Dec;70(6):1040-5. doi: 10.1093/ajcn/70.6.1040. PMID 10584049
- [Background] Kovacs EM, Lejeune MP, Nijs I, Westerterp-Plantenga MS. Effects of green tea on weight maintenance after body-weight loss. Br J Nutr. 2004 Mar;91(3):431-7. doi: 10.1079/BJN20041061. PMID 15005829
- [Background] Westerterp-Plantenga MS, Lejeune MP, Kovacs EM. Body weight loss and weight maintenance in relation to habitual caffeine intake and green tea supplementation. Obes Res. 2005 Jul;13(7):1195-204. doi: 10.1038/oby.2005.142. PMID 16076989
- [Derived] Gilardini L, Pasqualinotto L, Di Pierro F, Risso P, Invitti C. Effects of Greenselect Phytosome(R) on weight maintenance after weight loss in obese women: a randomized placebo-controlled study. BMC Complement Altern Med. 2016 Jul 22;16:233. doi: 10.1186/s12906-016-1214-x. PMID 27450231